CLINICAL TRIAL: NCT00259285
Title: Alimta (Pemetrexed) and Cisplatin Treatment as Neoadjuvant Therapy in Non Small Cell Lung Cancer
Brief Title: Pemetrexed and Cisplatin Treatment Before Surgery in Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was stopped early due to low enrollment.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9901; H3E-XM-S092
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-04

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2, intravenous (IV), every 21 days x 3 cycles
  Other Names: LY231514; Alimta
Drug: cisplatin — 75 mg/m2, intravenous (IV), every 21 days x 3 cycles

SUMMARY:
To determine the response to this regimen for therapy prior surgery in patients with locally advanced disease or metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-small-cell carcinoma of the lung
* Patients with locally advanced disease or metastatic disease, candidates to surgery after evaluation by oncologist and thoracic surgeon
* Tumour with possibility of curative surgery
* At least one uni-dimensionally measurable lesion
* Adequate pulmonary function to perform the planned surgical resection

Exclusion Criteria:

* Active infection (at the investigator's discretion)
* Pregnancy or breast-feeding
* Serious concomitant illness at the investigator's discretion
* Previous diagnosis of malignant disease
* They have received treatment during the last 30 days with a drug, other than the study drug, that has not received regulatory approval for any indication at the time of their entry in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM - 5 PM Eastern time (UTC/GMT- 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barakaldo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed + Cisplatin: Pemetrexed: 500 mg/m2, intravenous (IV), every 21 days x 3 cycles Cisplatin: 75 mg/m2, intravenous (IV), every 21 days x 3 cycles
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 61.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Spain | 10
Eastern Cooperative Oncology Group Functional Status [Number; unit: participants]
  0 - Fully Active | 8
  1 - Ambulatory, Restricted Strenuous Activity | 2
  2 - Ambulatory, No Work Activities | 0
  3 - Partially Confined to Bed, Limited Self Care | 0
  4 - Completely Disabled | 0
Race/Ethnicity [Number; unit: participants]
  Caucasian | 10
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meters] — weight divided by square height
  kilograms per square meters | 27.1 (4.3)
Corporal Surface (Body Surface Area) [Mean (Standard Deviation); unit: square meters] — The total surface area of the body (BSA). BSA was calculated by taking the square root of product of the weight in kilograms times the height in centimeters divided by 3600.
  square meters | 1.8 (0.2)
Height [Mean (Standard Deviation); unit: meters] | 1.6 (0.1)
Weight [Mean (Standard Deviation); unit: kilograms] | 72.8 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
Time Frame: every 21 day cycle (3 cycles) and 3-4 weeks after last cycle
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 10
participants
  Complete Response | 0
  Partial Response | 5
  Incomplete Response/Stable Disease | 4
  Progressive Disease | 1
  Not Evaluable | 0

2. Secondary Outcome: Pathologic Remissions After Surgery
Description: The status of the pathological response was evaluated on the basis of the original results of the histopathological examination of the tumour samples resected. A complete pathological response was defined as the absence of any viable tumour cell in the tumour samples obtained for histological examination.
Time Frame: surgical tumor resection (3-4 weeks after completing three 21-day cycles of therapy)
Population: 7 out of the 10 patients had surgery.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 7
participants
  Complete Remission - Yes | 5
  Complete Remission - No | 2

3. Secondary Outcome: Relapse-free Survival
Description: Results for this outcome measure were not analyzed because the trial stopped early due to low enrollment.
Time Frame: Every 21 day cycle (3 cycles) and then every 3 months for the first 2 years, every 6 months until 5 years have elapsed and annually thereafter
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 1
Other Adverse Events (participants affected / at risk) | 8
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Urinary tract infection (Infections and infestations) | 1/10 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 10% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Leukocytosis (Blood and lymphatic system disorders) | 1/10 (1)
Leukopenia (Blood and lymphatic system disorders) | 1/10 (1)
Neutrophilia (Blood and lymphatic system disorders) | 1/10 (1)
Abdominal Distension (Gastrointestinal disorders) | 1/10 (1)
Constipation (Gastrointestinal disorders) | 1/10 (1)
Diarrhoea (Gastrointestinal disorders) | 1/10 (1)
Nausea (Gastrointestinal disorders) | 4/10 (5)
Vomiting (Gastrointestinal disorders) | 2/10 (2)
Fatigue (General disorders) | 1/10 (1)
Mucosal inflammation (General disorders) | 1/10 (1)
Pyrexia (General disorders) | 1/10 (2)
Candidiasis (Infections and infestations) | 1/10 (1)
Respiratory tract infection (Infections and infestations) | 1/10 (1)
Alanine aminotransferase increased (Investigations) | 2/10 (2)
Aspartate aminotransferase increased (Investigations) | 2/10 (2)
Haemoglobin decreased (Investigations) | 1/10 (1)
Platelet count increased (Investigations) | 1/10 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1/10 (1)
Motor dysfunction (Nervous system disorders) | 1/10 (1)
Paraesthesia (Nervous system disorders) | 1/10 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3/10 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1/10 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1/10 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1/10 (1)
Rash (Skin and subcutaneous tissue disorders) | 2/10 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/10 (1)

LIMITATIONS AND CAVEATS:
Trial was stopped early due to low enrollment and the relapse-free survival outcome measure was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days